CLINICAL TRIAL: NCT04663841
Title: Mechanistic Circuit Markers of Transcranial Magnetic Stimulation Outcomes in Pharmacoresistant Depression
Brief Title: Neural Circuit Biomarkers of Transcranial Magnetic Stimulation Study
Status: Active, not recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency); Florida State University (Other); University of South Florida (Other); Medical University of South Carolina (Other); University of Minnesota (Other); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Brown University (Other); Providence VA Medical Center (U.S. Federal Agency); Dartmouth College (Other); Dartmouth-Hitchcock Medical Center (Other); White River Junction VA Medical Center (Unknown)
Responsible Party: Principal Investigator, Leanne Williams, Professor, Stanford University
Other Study IDs: 52695
Record Dates: First submitted 2020-11-27; First posted 2020-12-11 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: treatment resistant depression
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: transcranial magnetic stimulation — transcranial magnetic stimulation is delivered as part of routine care and is not managed by this observational study
  Other Names: TMS; repetitive transcranial magnetic stimulation

SUMMARY:
This study is currently recruiting Veterans only. The objective of this observational study is to test whether neuroimaging biomarkers of repetitive transcranial magnetic stimulation (TMS) can be prospectively replicated in a large ecologically valid sample. We focus on cognitive network connectivity as a predictive biomarker of the clinical effect of TMS, and as a response biomarker of change with TMS. We address this objective through a pragmatic approach in which we recruit patients undergoing routine clinical care and program evaluation in a Veterans Administration multi-site clinical TMS program.

DETAILED DESCRIPTION:
Although repetitive transcranial magnetic stimulation (TMS) is becoming a gold standard treatment for pharmacoresistant depression, we lack neural target biomarkers for identifying who is most likely to respond to TMS and why. To address this gap in knowledge this observational study evaluates neural targets defined by activation and functional connectivity of the dorsolateral prefrontal cortex-anchored cognitive control circuit, regions of the default mode network and attention circuit, and interactions with the subgenual anterior cingulate.

The study evaluates whether these targets and interactions between them change in a dose-dependent manner, whether changes in these neural targets correspond to changes in cognitive behavioral performance, and whether baseline and early change in neural target and cognitive behavioral performance predict subsequent symptom severity, suicidality, and quality of life outcomes.

This study is designed as a pragmatic, mechanistic observational trial partnering with the National Clinical TMS Program of the Veteran's Health Administration.

All veterans will receive a clinical course of TMS as part of their routine care. Those who agree to enrollment in the observational study will be assessed at 'baseline' prior to commencement of their TMS treatment, 'first week' after initiation of TMS (targeting five sessions) and 'post-treatment' at the completion of TMS (targeting 30 sessions).

Veterans will be assessed using functional magnetic resonance imaging (fMRI), a cognitive behavioral performance battery, and established questionnaires.

To our knowledge, our study will be the first pragmatic, mechanistic observational trial to use fMRI imaging and cognitive-behavioral performance as biomarkers of TMS treatment response in pharmacoresistant MDD.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years and older
* Meets Diagnostic and Statistical Manual edition 5 (DSM-5) criteria for Major Depressive Disorder (MDD) (as documented by the treating physician)
* Meet study criteria for pharmacoresistance in accordance with the Clinical transcranial magnetic stimulation (TMS) Program (i.e. failed at least one antidepressant in the current episode)
* Ability to obtain a motor threshold (MT) prior to the start of treatment
* Stable medical conditions and ability to maintain stability on current medication regimen for the duration of treatment
* Ability to participate in a daily treatment regimen
* Able to read, verbalize understanding, and voluntarily sign the Informed Consent Form prior to participating in any study-specific procedures or assessments

Exclusion Criteria:

* History of seizure disorder
* Structural or neurologic abnormalities present or in close proximity to the treatment site
* History of brain surgery
* Pacemaker or medical infusion device (unless magnetic resonance imaging compatible)
* History of traumatic brain injury within 60 days of the start of treatment
* Severe or uncontrolled alcohol or substance use disorders
* Active withdrawal from alcohol or substances
* Implanted device in the head
* Metal in the head
* Severe impediment to vision, hearing and/or hand movement, likely to interfere with ability to complete the assessments, or unable and/or unlikely to follow the study protocols
* Lifetime history of bipolar I disorder
* Inability to speak, read or understand English
* Plans to move out of the area during the study period
* Clinician and/or Investigator discretion for clinical safety or protocol adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with pharmacoresistant major depressive disorder (MDD) participating in the VA Clinical TMS Program. Given the complex nature of the veteran sample, the primary diagnosis of MDD may be comorbid with other disorders, including post-traumatic stress disorder (PTSD).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Go-NoGo elicited neural circuit function | Baseline
  Activation and connectivity assessed using functional magnetic resonance imaging during a GoNoGo task
Go-NoGo elicited neural circuit function | Up to 2 weeks
  Activation and connectivity assessed using functional magnetic resonance imaging during a GoNoGo task
Go-NoGo elicited neural circuit function | Up to 8 weeks
  Activation and connectivity assessed using functional magnetic resonance imaging during a GoNoGo task
N-Back elicited neural circuit function | Baseline
  Activation and connectivity assessed using functional magnetic resonance imaging during an N-Back task
N-Back elicited neural circuit function | Up to 2 weeks
  Activation and connectivity assessed using functional magnetic resonance imaging during an N-Back task
N-Back elicited neural circuit function | Up to 8 weeks
  Activation and connectivity assessed using functional magnetic resonance imaging during an N-Back task
Resting state neural circuit function | Baseline
  connectivity assessed using functional magnetic resonance imaging during a resting condition
Resting state neural circuit function | Up to 2 weeks
  connectivity assessed using functional magnetic resonance imaging during a resting condition
Resting state neural circuit function | Up to 8 weeks
  connectivity assessed using functional magnetic resonance imaging during a resting condition

SECONDARY OUTCOMES:
Symbol Digit Coding Test | Baseline
  Cognitive-Behavioral Performance accuracy on the Symbol Digit Coding Test
Symbol Digit Coding Test | Up to 2 weeks
  Cognitive-Behavioral Performance accuracy on the Symbol Digit Coding Test
Symbol Digit Coding Test | Up to 8 weeks
  Cognitive-Behavioral Performance accuracy on the Symbol Digit Coding Test
Stroop Test | Baseline
  Cognitive-Behavioral Performance accuracy and reaction time on the Stroop Test
Stroop Test | Up to 2 weeks
  Cognitive-Behavioral Performance accuracy and reaction time on the Stroop Test
Stroop Test | Up to 8 weeks
  Cognitive-Behavioral Performance accuracy and reaction time on the Stroop Test
Shifting Attention Test | Baseline
  Cognitive-Behavioral Performance accuracy and reaction time on the Shifting Attention Test
Shifting Attention Test | Up to 2 weeks
  Cognitive-Behavioral Performance accuracy and reaction time on the Shifting Attention Test
Shifting Attention Test | Up to 8 weeks
  Cognitive-Behavioral Performance accuracy and reaction time on the Shifting Attention Test
Continuous Performance Test | Baseline
  Cognitive-Behavioral Performance accuracy and reaction time on the Continuous Performance Test platform
Continuous Performance Test | Up to 2 weeks
  Cognitive-Behavioral Performance accuracy and reaction time on the Continuous Performance Test platform
Continuous Performance Test | Up to 8 weeks
  Cognitive-Behavioral Performance accuracy and reaction time on the Continuous Performance Test platform
Depressive Symptoms | Baseline
  Clinical outcome assessed using the Quick Inventory of Depressive Symptoms (QIDS)- Self Report Form. The total score ranges from 0 to 27 with higher scores indicating greater severity.
Depressive Symptoms | Up to 2 weeks
  Clinical outcome assessed using the Quick Inventory of Depressive Symptoms (QIDS)- Self Report Form. The total score ranges from 0 to 27 with higher scores indicating greater severity.
Depressive Symptoms | Up to 8 weeks
  Clinical outcome assessed using the Quick Inventory of Depressive Symptoms (QIDS)- Self Report Form. The total score ranges from 0 to 27 with higher scores indicating greater severity.
Daily function related to quality of life | Baseline
  Clinical outcome assessed using the Veterans' RAND 36-item Health Survey (VR-36). All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible.
Daily function related to quality of life | Up to 2 weeks
  Clinical outcome assessed using the Veterans' RAND 36-item Health Survey (VR-36). All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible.
Daily function related to quality of life | Up to 8 weeks
  Clinical outcome assessed using the Veterans' RAND 36-item Health Survey (VR-36). All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible.
Suicidal ideation | Baseline
  Columbia-Suicide Severity Rating Scale (C-SSRS). The total score ranges from 2 to 25, with a higher number indicating more intense ideation and greater risk.
Suicidal ideation | Up to 2 weeks
  Columbia-Suicide Severity Rating Scale (C-SSRS). The total score ranges from 2 to 25, with a higher number indicating more intense ideation and greater risk.
Suicidal ideation | Up to 8 weeks
  Columbia-Suicide Severity Rating Scale (C-SSRS). The total score ranges from 2 to 25, with a higher number indicating more intense ideation and greater risk.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Williams, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Department of Psychiatry, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No